CLINICAL TRIAL: NCT06975891
Title: Subjective and Objective Performance of Systane PRO Versus Refresh Optive Mega-3 in Dry Eye Patients
Brief Title: Performance of Systane PRO Versus Refresh Optive Mega-3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Scripps Poway Eyecare and Optometry (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: JM-25-01
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Systane PRO then Refresh Optive Mega-3 (Other)
  Interventions: Drug: Systane PRO; Drug: Refresh Optive MEGA-3
- Refresh Optive Mega-3 then Systane PRO (Other)
  Interventions: Drug: Systane PRO; Drug: Refresh Optive MEGA-3

INTERVENTIONS:
Drug: Systane PRO — Lubricating Eyedrops
Drug: Refresh Optive MEGA-3 — Lubricating Eyedrops

SUMMARY:
Single site, prospective, double-masked, randomized-controlled, cross-over study of the subjective and objective performance of 2 different eyedrops. Subjects will be assessed at a screening visit, and 3 follow-up visits. Clinical evaluations will include patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who currently have moderate symptoms of dry eye as defined by a baseline OSDI score of 23-32 inclusive.
* Subjects between ages of 18-65 inclusive.
* Subjects who do not currently wear contact lenses.
* Subjects willing to fill out a daily diary during the duration of the study.
* Subjects willing to comply with the prescribed regimen and schedule of eye drops.
* Subjects willing to attend all study visits.

Exclusion Criteria:

* Have an ophthalmologic diagnosis of: allergy, viral or bacterial conjunctivitis, anterior blepharitis, parasitic infestations in any ocular structure or its adnexa, unresolved ocular trauma, ocular surface scarring diseases, corneal or conjunctival ulcers, filamentous keratitis, neurotrophic keratitis, bulous keratopathy, neoplastic diseases on the ocular surface or adnexa, diseases with fibrovascular proliferations on the conjunctival and/or corneal surface, retinal and/or posterior diseases that require treatment or threaten the visual prognosis, or glaucoma.
* Eyelid disorders that cause eyelid malposition, limit adequate eyelid closure or opening or cause epiphora.
* History of herpetic keratitis or ocular surgery.
* Have dry eye management that requires the implementation of any treatments (except artificial tears) of stage 2 of the recommendations in the treatment and management by stages for the dry eye disease of the TFOS DEWS I| (Tear Film and Ocular Surface Society Dry Eye Workshop I).
* Have a history of drug addiction or drug dependence currently or within the last two years before signing the ICF.
* Have another medical condition, acute or chronic, that in the opinion of the investigator could increase the risk associated with participation in the study or the administration of the investigational product, or that could interfere with the interpretation of the results of the study.
* Pregnant or lactating.
* Current use of contact lenses.
* Have participated in another clinical research study ≤30 days before screening visit.
* Any use of eye drops, whether OTC or Rx, in last 14 days.
* Subjects who have previously used either investigational product in the past.
* Have known hypersensitivity to the components of the investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
OSDI Questionnaire | Change from baseline to 28 days
  The OSDI© is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. The OSDI© is a valid and reliable instrument for measuring dry eye disease (normal, mild to moderate, and severe) and effect on vision-related function.

SECONDARY OUTCOMES:
Visual Analog Score | Change from baseline to 28 days
  Subjects are asked to draw a vertical line on the scale below to best describe how they have felt about eye comfort for the past 4 weeks. Scale is from 0 to 100 with 0 representing no discomfort and 100 representing max discomfort.

OTHER OUTCOMES:
Likert Questionnaire | 28 days after start of eyedrop
  Subjects are asked to rate how likely they would be to recommend these eyedrops for the treatment of dry eye symptoms: Very Unlikely, Somewhat Unlikely, Neither Likely nor Unlikely, Somewhat Likely, Very Likely.
Eyedrop preference question | 28 days after start of second eyedrop
  Subjects are asked to select which drop they felt did a better job relieving dry eye symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mashouf, OD, Principal Investigator — Scripps Optometric Group
Locations (1):
- Scripps Poway Eyecare & Optometry, San Diego, California, United States